CLINICAL TRIAL: NCT02183545
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 1060469 in Healthy Asian Male Volunteers in a Randomized, Double-blind, Placebo-controlled Design
Brief Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 1060469 in Healthy Asian Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1333.3
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- BI 1060469 (Experimental): single rising doses given as tablet
  Interventions: Drug: BI 1060469
- Placebo (Placebo Comparator): given as tablet (matching placebo of BI 1060469)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1060469 — single rising doses given as tablet
  Arms: BI 1060469
Drug: Placebo — given as tablet (matching placebo of BI 1060469)
  Arms: Placebo

SUMMARY:
The objective of this single rising dose study (SRD) is to investigate safety, tolerability, and pharmacokinetics of single rising doses of BI 1060469 in healthy Asian male subjects.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males based upon a complete medical history, including a physical examination, vital signs (blood pressure, pulse rate), 12-lead ECG, and clinical laboratory tests
2. Chinese ethnicity, Japanese ethnicity according to the following criteria:

   Chinese; born in China or ethnic Chinese born outside of China, and a descendent of 4 ethnic Chinese grandparents who were all born in china Japanese; born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who were all born in Japan
3. Age within the range of 18 to 45 years
4. Body mass index within the range of 18.5 and 25 kg/m2
5. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice(GCP) and local legislation.

Exclusion criteria:

1. Any finding in the medical examination (including blood pressure, pulse rate or ECG(electrocardiogram)) deviating from normal and judged clinically relevant by the investigator. Pulse rate outside the range of 50-90 beat per minute or blood pressure outside the ranges of 90-140 for systolic and 50-90 mmHg for diastolic blood pressure if confirmed by repeat measurement.
2. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
3. Serum creatinine laboratory value outside the normal range
4. Glomerular Filtration Rate according to CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) Formula < 60 ml/ min
5. Current or history of relevant kidney, urinary tract diseases or abnormalities (i.e. nephrolithiasis, hydronephrosis, acute or chronic nephritis, renal injury, renal failure, infections)
6. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
7. Surgery of the gastrointestinal tract that could interfere with kinetics of the study drug
8. Diseases of the central nervous system (such as epilepsy), central neurological disorders or psychiatric disorders
9. History of relevant orthostatic hypotension, fainting spells, or blackouts
10. Relevant chronic or acute infections
11. History of relevant allergy/hypersensitivity (including allergy to the trial medication or its excipients)
12. Intake of drugs with a long half-life (greater than 24 hours) within 30 days or less than 10 half-lives of the respective drug prior to study drug administration
13. Intake of any NSAIDs(Nonsteroidal anti-inflammatory drugs), COX2(Cyclooxygenase-2) inhibitors, aspirin, ACE(Angiotensin Converting Enzyme) inhibitors, H2-blockers or OTC(Over the Counter Drug)- or nutripharmaceuticals between screening examination and drug administration
14. Use of drugs that might reasonably influence the results of the trial (including renal function measurements) or that might prolong the QT/QTc interval within 14 days prior to study drug administration
15. Participation in another trial with investigational drug administration within 60 days prior to administration of trial medication
16. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes/day)
17. Inability to refrain from smoking on specified trial days
18. Alcohol abuse (consumption of more than 30 g/day)
19. Drug abuse or positive drug screen
20. Blood donation (more than 100 mL within 30 days prior to administration of trial medication or intended during the trial)
21. Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
22. Inability to comply with dietary regimen of trial site
23. A marked baseline prolongation of QT/QTc interval (such as repeated demonstration of a QTc interval greater than 450 ms) or any other relevant ECG finding
24. A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
25. Subject is assessed by the investigator as unsuitable for inclusion, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
number of subjects with drug-related adverse events | up to 14 days after drug administration

SECONDARY OUTCOMES:
Maximum concentration of BI 1060469 (Cmax) | up to 72 hours after drug administration
Area Under the concentration-time curve of BI 1060469 over time interval from 0 interpolated to infinity ((AUC0-infinity) | up to 72 hours after drug administration
Area Under the concentration-time curve of BI 1060469 (AUC0- tz) | up to 72 hours after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- South Korea (2):
  - 1333.3.82002 Boehringer Ingelheim Investigational Site, Busan
  - 1333.3.82001 Boehringer Ingelheim Investigational Site, Seoul